CLINICAL TRIAL: NCT03053193
Title: MammaPrint, BluePrint, and Full-genome Data Linked With Clinical Data to Evaluate New Gene EXpression Profiles: An Adaptable Registry (FLEX)
Brief Title: MammaPrint, BluePrint, and Full-genome Data Linked With Clinical Data to Evaluate New Gene EXpression Profiles
Acronym: FLEX
Status: Recruiting | Type: Observational
Sponsor: Agendia (Industry)
Responsible Party: Sponsor
Other Study IDs: FLEX Registry
Record Dates: First submitted 2017-02-09; First posted 2017-02-15 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: breast cancer; stage I; stage II; stage III
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Tumor tissue acquired as part of a standard of care biopsy or surgical procedure will be sent to Agendia for testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MammaPrint and BluePrint testing: All patients will receive MammaPrint and BluePrint testing using the full-genome testing data chip. Treatment will be at the discretion of the physician while adhering to NCCN guidelines.
  Interventions: Diagnostic Test: MammaPrint, BluePrint, and Full-Genome Testing

INTERVENTIONS:
Diagnostic Test: MammaPrint, BluePrint, and Full-Genome Testing — Agendia will run MammaPrint and BluePrint tests using the full genome testing array.
  Other Names: MammaPrint, BluePrint

SUMMARY:
The FLEX Registry will be implemented to operate as a large-scale, population based, prospective registry. All patients with stage I to III breast cancer who receive MammaPrint® and BluePrint testing on a primary breast tumor are eligible for entry into the FLEX Registry, which is intended to enable additional study arms at low incremental effort and cost. FLEX Registry will utilize an adaptive design, where additional targeted substudies and arms can be added after the initial study is opened.

DETAILED DESCRIPTION:
The FLEX Registry will include all patients with stage I-III breast cancer who have received MammaPrint and BluePrint testing in any clinical setting. Study arm appendices will specify treatment arm, inclusion criteria, and number of patients needed. Approximately 30,000 patients from 125+ US based institutions will be enrolled.

Treatment is at the discretion of the physician adhering to NCCN approved regimens of a recognized alternative.

Clinical data will be collected and entered online at the time points listed: patient enrollment, time of treatment, 1 year post-treatment, and 3, 5, and 10 years post diagnosis.

Objectives:

* Create a large scale, population-based registry of full genome expression data and clinical data to investigate new gene associations with prognostic and/or predictive value
* Utilize shared registry infrastructure to examine smaller groups of interest
* Generate hypotheses for targeted subset analyses and trials based on full genome data

FLEX is an observational (phase IV) study.

ELIGIBILITY:
Inclusion Criteria:

* Stage I, II, or III patients who receive MammaPrint, with or without BluePrint testing (male or female)
* Informed consent form signed on the same day or before enrollment
* New primary lesion

Exclusion Criteria:

* Tumor sample shipped to Agendia with ≤ 30% tumor cells or that fails QA or QC criteria
* Metastatic disease
* Recurrent disease
* Stage 0 disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include patients with stage I, II, or III breast cancer that have signed an informed consent, and are eligible to receive chemotherapy and endocrine therapy. Patients will be excluded if they have metastatic disease or do not have ample tissue to send to Agendia for testing.
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2017-04-28 (Actual); Primary Completion 2037-04 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
A large scale registry of full genome expression data to investigate new gene associations with prognostic and/or predictive value will be created. | 10 years
  Create a large scale registry of full genome expression data with clinical data to investigate possible new gene associations with prognostic or predictive value.
A shared registry infrastructure to examine smaller groups of interest. | 10 years
  Create a shared registry infrastructure to examine smaller groups of interest.

SECONDARY OUTCOMES:
Subset analyses based on full genome data will be created. | 10 years
  Use full genome data to analyze subsets.

CONTACTS AND LOCATIONS:
Overall Officials: William Audeh, MD, Study Director — Agendia, Inc.; Joyce O'Shaughnessy, MD, Principal Investigator — Texas Oncology - Baylor Charles A. Sammons Center
Locations (134):
- United States (130):
  - CHS Grandview, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Arizona Oncology Associates, PC, Phoenix, Arizona
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Adventist Health - Bakersfield, Bakersfield, California
  - Comprehensive Cancer Center at Desert Regional Medical Center, Palm Springs, California
  - North Valley Breast Clinic, Redding, California
  - UCSF Breast Care Center, San Francisco, California
  - Valley Breast Care, Van Nuys, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - University of Colorado Cancer Center, Aurora, Colorado
  - Comprehensive Breast Care of Denver, Denver, Colorado
  - Rocky Mountain Cancer Center - Lakewood, Lakewood, Colorado
  - Vail Health - Shaw Cancer Center, Vail, Colorado
  - St. Mary's Hospital, Waterbury, Connecticut
  - Medical Oncology and Hematology Consultants, Newark, Delaware
  - Breast Specialists of South Florida, Atlantis, Florida
  - JFK Medical Center, Atlantis, Florida
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Morton Plant Hospital, Clearwater, Florida
  - Halifax Health - Center for Oncology, Daytona Beach, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - St. Vincent Hospital / Mayo Clinic, Jacksonville, Florida
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - Sylvester Comprehensive Cancer Center - University of Miami, Miami, Florida
  - Miami Cancer Institute at Baptist Health, Inc, Miami, Florida
  - Cancer Care Centers of Brevard, Rockledge, Florida
  - St. Joseph's Hospital - Baycare, Tampa, Florida
  - University of South Florida, Tampa, Florida
  - Winter Haven Hospital, Winter Haven, Florida
  - Phoebe Health, Albany, Georgia
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Emory University - Winship Cancer Institute, Atlanta, Georgia
  - Southeast Georgia Health System - Physician Associates, Brunswick, Georgia
  - DeKalb Medical Center, Decatur, Georgia
  - Candler Hospital, Savannah, Georgia
  - Tift Regional Health System, Tifton, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Saint Alexius Medical Center, Hoffman Estates, Illinois
  - Affiliated Oncologists, Oak Lawn, Illinois
  - Parkview Health, Fort Wayne, Indiana
  - Louisiana State University, Shreveport, Louisiana
  - Northern Light Breast Care, Portland, Maine
  - Luminis Health Center for Cancer & Blood Disorders, Annapolis, Maryland
  - Mercy Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Maryland Oncology Hematology - Bethesda, Bethesda, Maryland
  - Maryland Oncology Hematology - Brandywine, Brandywine, Maryland
  - Maryland Oncology Hematology - Clinton, Clinton, Maryland
  - Maryland Oncology Hematology, PA, Columbia, Maryland
  - UPMC at Western Maryland Health System, Cumberland, Maryland
  - Frederick Oncology Hematology Associates, Frederick, Maryland
  - Maryland Oncology Hematology - Aquilino Cancer Center, Rockville, Maryland
  - Maryland Oncology Hematology, PA, Silver Spring, Maryland
  - Mercy Medical Center, Springfield, Massachusetts
  - St. John Hospital, Grosse Pointe Woods, Michigan
  - Sparrow Cancer Center, Lansing, Michigan
  - Beaumont Breast Care Center, Royal Oak, Michigan
  - Providence - Providence Park Hospital, Southfield, Michigan
  - Comprehensive Breast Care, Troy, Michigan
  - Minnesota Oncology, Minneapolis, Minnesota
  - Boone Hospital Center, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - New York Oncology Hematology, Albany, New York
  - Broome Oncology, Binghamton, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Lake Success Oncology / ProHealth Care, Lake Success, New York
  - NYU Winthrop Hospital, Mineola, New York
  - Northwell Health- Northern Westchester Hospital, Mount Kisco, New York
  - Kings County Hospital, New York, New York
  - Hematology Oncology Center of Rockland at Nyack, Nyack, New York
  - University of Rochester - Pluta Cancer Center, Rochester, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Northwell Health- Phelps Hospital, Tarrytown, New York
  - Akron General Medical Center, Akron, Ohio
  - TriHealth Cancer Institutes, Cincinnati, Ohio
  - Oncology Hematology Care, Cincinnati, Ohio
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Legacy Good Samaritan Medical Center, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - St. Luke's Hospital, Bethlehem, Pennsylvania
  - Consultants in Medical Oncology and Hematology, P.C., Broomall, Pennsylvania
  - Alliance Cancer Specialists, Horsham, Pennsylvania
  - St. Mary Medical Center, Langhorne, Pennsylvania
  - Allegheny Health Network, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Centers, Pittsburgh, Pennsylvania
  - Grandview Hospital, Sellersville, Pennsylvania
  - Roper St. Francis Physician Partners - Breast Surgery, Charleston, South Carolina
  - Tidelands Health Coastal Carolina Breast Center, Georgetown, South Carolina
  - West Cancer Center, Germantown, Tennessee
  - Nashville Breast Center, Nashville, Tennessee
  - Texas Oncology - Allen, Allen, Texas
  - Harrington Cancer Center, Amarillo, Texas
  - Texas Oncology - Austin, Austin, Texas
  - Texas Oncology - Bedford, Bedford, Texas
  - Texas Oncology - Carrollton, Carrollton, Texas
  - CHRISTUS Spohn Cancer Center, Corpus Christi, Texas
  - Texas Oncology - Methodist Dallas Cancer Center, Dallas, Texas
  - Texas Oncology - Presbyterian, Dallas, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Denton, Denton, Texas
  - Texas Oncology - Flower Mound, Flower Mound, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Texas Oncology - Grapevine, Grapevine, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - Texas Oncology Willowbrook, Houston, Texas
  - Oncology Consultants, Katy, Texas
  - University of Texas Medical Branch, League City, Texas
  - Texas Oncology - Longview, Longview, Texas
  - Texas Tech UHSC - Southwest Cancer Center, Lubbock, Texas
  - Texas Oncology - McKinney, McKinney, Texas
  - Texas Oncology - Plano East, Plano, Texas
  - Texas Oncology - Plano West, Plano, Texas
  - Texas Oncology, PA - Metropolitan, San Antonio, Texas
  - Texas Oncology, PA - Northeast, San Antonio, Texas
  - UT Health Cancer Center, San Antonio, Texas
  - Texas Oncology PA -San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology, PA - Stone Oak, San Antonio, Texas
  - Texas Oncology - Sugar Land, Sugar Land, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Texas Oncology - Waco, Waco, Texas
  - Texas Oncology - Webster, Webster, Texas
  - Ogden Regional Cancer Center, Ogden, Utah
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Columbia St. Mary's, Milwaukee, Wisconsin
- Canada (2):
  - William Osler Cancer Centre, Brampton, Ontario
  - Thunder Bay Regional Health Sciences Centre, Thunder Bay, Ontario
- University General Hospital Alexandra, Athens, Greece
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brufsky AM, Hoskins KF, Conter HJ, Kelemen P, Habibi M, Samian L, Rahman RL, Lee L, Dias EC, Hampton R, Sieling BA, Osborne CR, Brown E, Elayoubi JA, Sharma P, Ramadurai J, Matt-Amaral L, Santillan AA, Davis S, Albaneze P, Ramaswamy H, Chmielewski-Stivers N, Menicucci A, Audeh W, Whitworth P, Johnson N, O'Shaughnessy J. MammaPrint predicts chemotherapy benefit in HR+HER2- early breast cancer: FLEX Registry real-world data. JNCI Cancer Spectr. 2025 Sep 1;9(5):pkaf079. doi: 10.1093/jncics/pkaf079. PMID 40796181